CLINICAL TRIAL: NCT07253090
Title: The Comparative Study on the Alteration of Endoscopic Ultrasound Guided Portal Pressure Gradient in Esophageal Varices After Ligation and Sclerotherapy
Brief Title: EUS-PPG Alteration After Ligation and Sclerotherapy in Esophageal Varices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-0708
Record Dates: First submitted 2025-11-17; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-07

CONDITIONS: Esophagogastric Varices
MeSH Terms: interventions — Sclerotherapy; Ligation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-PPG alteration in esophageal varices after ligation (Other)
  Interventions: Procedure: Ligation for esophageal varices
- EUS-PPG alteration in esophageal varices after sclerotherapy (Experimental)
  Interventions: Procedure: Sclerotherapy for esophageal varices

INTERVENTIONS:
Procedure: Sclerotherapy for esophageal varices — EUS-PPG alteration in esophageal varices after sclerotherapy
  Arms: EUS-PPG alteration in esophageal varices after sclerotherapy
Procedure: Ligation for esophageal varices — EUS-PPG alteration in esophageal varices after Ligation
  Arms: EUS-PPG alteration in esophageal varices after ligation

SUMMARY:
Acute variceal bleeding due to cirrhotic portal hypertension is a life-threatening emergency in gastroenterology. Current preventive strategies include non-selective β-blockers (e.g., carvedilol/propranolol), endoscopic therapy (sclerotherapy or band ligation), and transjugular intrahepatic portosystemic shunt (TIPS). While pharmacological and TIPS interventions directly reduce portal pressure, the impact of endoscopic therapies on portal hemodynamics remains controversial. The hepatic venous pressure gradient (HVPG), measured via transjugular catheterization as the difference between wedged and free hepatic venous pressures, is the gold standard for assessing portal pressure. Clinically significant portal hypertension (CSPH) is defined as HVPG ≥10 mmHg, with values >12 mmHg predicting variceal formation and bleeding risk.

Traditional views suggest that non-selective β-blockers and transjugular intrahepatic portosystemic shunt (TIPS) can reduce portal vein pressure. Does endoscopic intervention affect portal vein pressure? Previous studies have explored changes in HVPG in the acute phase after esophageal variceal sclerotherapy and ligation therapy, with inconsistent results. In the study by Toyonaga et al., HVPG was rechecked 2 weeks after sclerotherapy, and the average decreased from 17.9 mmHg to 17.6 mmHg (J Hepatol. 1994 Oct;21(4):515-20). In the study by Gonzalo Bada et al., HVPG values increased from 16.5 mmHg to 19.5 mmHg on average 24 hours after ligation therapy (Rev Esp Enferm Dig. 2020 Jun;112(6):456-461). However, in a prospective randomized controlled study conducted by Avgerinos et al., which compared changes in HVPG within 5 days after ligation and sclerotherapy, and found that HVPG significantly increased after sclerotherapy, while there was no significant change in HVPG after ligation (Hepatology. 2004 Jun;39(6):1623-30).

The investigators speculate that the inconsistent results mentioned above may be related to the limitations of HVPG, which inaccurately reflects pre-sinusoidal/extrahepatic portal hypertension and is influenced by technical factors (e.g., catheter position, sedation). Emerging evidence suggests endoscopic ultrasound-guided portal pressure gradient (EUS-PPG) measurement may overcome these limitations. Recent studies demonstrate strong correlations between EUS-PPG and HVPG, as well as associations with variceal severity and Child-Pugh class. However, data on chronic portal pressure changes (≥3 months) post-endoscopic therapy are lacking.

This prospective study aims to evaluate chronic changes in EUS-PPG 3-6 months after endoscopic variceal ligation (EVL) or sclerotherapy in cirrhotic patients receiving primary/secondary prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

Cirrhotic patients admitted for primary/secondary prevention due to esophageal and gastric varices, and willing to sign the informed consent form.

Exclusion Criteria:

1. Refusing to sign the informed consent form;
2. Age < 18 years, or ≥ 81 years;
3. Coagulopathy (INR > 1.5);
4. Markedly decreased platelets (<20,000/μL);
5. Propranolol/carvedilol was used 24h before admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The altered value of portal vein pressure gradient measured under EUS after sclerotherapy or ligation for esophegeal varices | 3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China